CLINICAL TRIAL: NCT03724721
Title: To Investigate the Safety and Efficacy of Vacuum Bottle Plus Catheter for Drainage of Pneumothorax
Brief Title: Pneumothorax Drainage With Vacuum Bottle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201805105DINA
Record Dates: First submitted 2018-10-16; First posted 2018-10-30 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Iatrogenic Pneumothorax; Vacuum Bottle Assisted Needle Aspiration
Keywords: Pneumothorax/therapy; Drainage
MeSH Terms: conditions — Pneumothorax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pneumothorax drainage (Experimental): Pneumothorax drainage with vacuum bottle plus intercostal catheter
  Interventions: Procedure: vacuum bottle

INTERVENTIONS:
Procedure: vacuum bottle — using vacuum bottle plus catheter for drainage of pneumothorax

SUMMARY:
The use of vacuum bottle in drainage of pneumothorax was seldom reported. This study aims to investigate the safety of vacuum bottle plus non-tunneled catheter for drainage of iatrogenic pneumothorax.

DETAILED DESCRIPTION:
For aspiration or drainage of pneumothorax, a 16-gauge or 18-gauge over-the-needle non-tunneled catheter, a pigtail, or chest tube are frequently used to penetrate the pleural space. A 50-ml or 60-ml syringe may be connected to the over-the-needle catheter or a pigtail for simple aspiration, while underwater-sealed bottle or suction drainage connected to chest tube for drainage of pneumothorax. Vacuum bottle for removing pleural effusion are frequently reported in literature and common in daily practice. However, the use of vacuum bottle in drainage of pneumothorax was seldom reported. This study aims to investigate the safety of vacuum bottle plus non-tunneled catheter for drainage of iatrogenic pneumothorax.

ELIGIBILITY:
1. Inclusion criteria:

   · Clinical diagnosis of pneumothorax
2. Exclusion criteria

   * Bleeding tendency
   * Tension pneumothorax
   * Shock

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-08-23 (Actual); Primary Completion 2020-02-11 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Intrapleural pressure during vacuum bottle air drainage | Within 1 hour
  The investigator will measure the intrapleural pressure during air drainage at 5 seconds, 10 seconds, 15 seconds, 20 seconds, 25 seconds, 30 seconds, 1 minute, 2 minutes, 5 minutes, 10 minutes, 15 minutes and until finished (the remaining with 5 minutes interval). It is proposed in previous studies that it is safe if the intrapleural pressure is less than 20 cmH2O during the procedure.

SECONDARY OUTCOMES:
Rate of reexpansion pulmonary edema | within 1day after the procedure
  By calculating the rate of reexpansion pulmonary edema among vacuum bottle assisted drainage can investigator determine whether it is a safe procedure
The resolution rate of pneumothorax | 1 week
  Chest X ray will be taken after the procedure and compared with that taken before the procedure. By using Rhea method, the investigator can compare the percentage of remaining pneumothorax compared with that before the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Kuo Yao-Wen, MD, Principal Investigator — National Taiwan University Hospital; Chen Shih-Yu, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Chen SY, Kuo YW, Ho CC, Wu HD, Wang HC. Safety and efficacy of vacuum bottle plus catheter for drainage of iatrogenic pneumothorax. BMC Pulm Med. 2022 Jun 7;22(1):221. doi: 10.1186/s12890-022-02009-8. PMID 35672758